CLINICAL TRIAL: NCT01165619
Title: Detailed Clinical, Biochemical and Genetic Characterization in GnRH Deficiency Disorders
Brief Title: Detailed Clinical, Biochemical and Genetic Characterization in Gonadotropin-releasing Hormone (GnRH) Deficiency Disorders
Status: Terminated | Type: Observational
Why Stopped: the Principal Investigator left the institution
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Nelly Pitteloud, MD, Massachusetts General Hospital
Other Study IDs: 1200204347-BL
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Idiopathic Hypogonadotropic Hypogonadism; Hypothalamic Amenorrhea
MeSH Terms: conditions — Idiopathic Hypogonadotropic Hypogonadism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, plasma, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Hypothalamic Amenorrhea: This group is for pre-menopausal women between the aged 18-40 who have been previously diagnosed with Hypothalamic Amenorrhea. They can be currently diagnosed or may have recovered.
- Healthy Adult Men: This group is men over the age of 18 who do not have any history of reproductive disorders or chronic disease.
- Healthy Adult Women: This group is pre-menopausal, regularly menstruating women ages 18-40 who do not have a history of reproductive disorders or chronic disease.
- Idiopathic Hypogonadotropic Hypogonadism: This group is for adult men and women over the age of 18 who have been diagnosed with Idiopathic Hypogonadotropic Hypogonadism with or without anosmia.

SUMMARY:
In this study, we will measure levels of reproductive hormones and metabolic markers in subjects with isolated GnRH deficiency disorders and compare them to healthy control populations. Our goals are (1) to chart the range of hormonal and metabolic biomarkers in healthy subjects and those with reproductive disorders and (2) to correlate reproductive and metabolic phenotypes with genetic changes within patients with reproductive disorders and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 for men
* Between the ages of 18 and 40 for women
* For reproductive disorder population: Current or previous diagnosis of Idiopathic Hypogonadotropic Hypogonadism or Hypothalamic Amenorrhea

Exclusion Criteria:

* chronic disease (hypertension, high cholesterol, diabetes, asthma, etc)
* polycystic ovarian syndrome for women
* prescription medication use (other than allergy meds) for control populations
* irregular menstrual cycles for healthy female control population (cycle length longer than 35 days or shorter than 25 days. cycle length varies by more than 5 days. less than 9 periods per year)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The reproductive disorder populations will be recruited from the reproductive endocrine clinic at the Mass General Hospital. The control populations will be recruited from Boston and surrounding communities
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Serum/plasma markers | baseline
  At the study visit, serum and plasma samples will be taken to measure levels of reproductive hormones and metabolic markers in the subjects' blood.

SECONDARY OUTCOMES:
Genetics | baseline
  At the study visit, blood will be taken and DNA cell lines will be made to screen for genes that potentially contribute to the development of reproductive disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States